CLINICAL TRIAL: NCT01286129
Title: Comparative Responses to Nasal Allergen Challenge in Allergic Rhinitic Subjects With or Without Asthma
Brief Title: Nasal Allergen Challenge in Rhinitic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: AllerGen NCE Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FP-2005-3; CER1223 (Other: Ethics committee)
Record Dates: First submitted 2011-01-13; First posted 2011-01-31 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergic asthmatic (Active Comparator): Subjects with allergic asthma will undergo nasal allergen provocations with either house dust mite or cat pelt.
  Interventions: Procedure: Nasal allergen challenge
- Allergic rhinitic without asthma (Active Comparator): Subjects with allergic rhinitis without asthma will undergo nasal allergen provocations with either house dust mite or cat pelt.
  Interventions: Procedure: Nasal allergen challenge

INTERVENTIONS:
Procedure: Nasal allergen challenge — Allergen sprayed into nostrils. Allergen used will be house dust mite or cat allergen. Allergens will be given in increasing ten-fold dilutions until a positive response occurs.

SUMMARY:
Background: Nasal allergen challenge (NAC) is useful to study the pathophysiology of rhinitis, and multiple challenges may more adequately approximate natural exposure.

Objective: To determine the effect of 4 consecutive daily NAC, on clinical and inflammatory parameters in rhinitics with or without asthma.

DETAILED DESCRIPTION:
The study will be performed outside the pollen season. On a baseline visit, 2 to 7 days prior to control challenge, allergy skin prick tests and methacholine inhalation test will be done. Prior to first allergen challenge, skin titration will be done using tenfold dilutions of the allergen chosen for nasal challenges. Subsequent to baseline visit, a control challenge will be done, followed, a week later, by repeated NACs. NACs will be done over 4 consecutive days, in the morning. Nasal peak inspiratory flows (NPIF), oral peak expiratory flows (PEF), and symptoms will be recorded at baseline and at regular intervals over 7 hours post-challenge on each challenge day. Induced sputum and nasal lavage specimen will be obtained 7 hours following the control challenge and the first and last NAC.

ELIGIBILITY:
Inclusion Criteria:

* To have a positive reaction to one or more allergen on prick tests.
* Non smokers
* No respiratory track infection for at least one month prior to the study.
* Positive reaction to cat hair and/or house dust mite (Dermatophagoides pteronyssinus) aeroallergens on allergy skin prick tests and report rhinitis symptoms when exposed to an environment containing this allergen.
* Asthmatic subjects using only inhaled beta-2 agonists on an as needed basis for their asthma treatment.
* Asthmatic subjects with a history of asthma of at least 6 months.
* Asthmatic subjects with PC20 methacholine lower or equal to 8 mg/ml.
* Allergic rhinitic subjects never experienced any asthma symptoms or took any asthma medication in the past.
* Allergic rhinitic subjects with a provocative concentration of methacholine (PC20 higher than 16 mg/ml.

Exclusion Criteria:

* Smokers or ex smokers less than 6 months or more than 10 pack-years.
* Asthmatic subjects using or used in the past 3 months inhaled or oral corticosteroids.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Rousseau MC, Boulay ME, Goronfolah L, Denburg J, Keith P, Boulet LP. Comparative responses to nasal allergen challenge in allergic rhinitic subjects with or without asthma. Allergy Asthma Clin Immunol. 2011 Apr 20;7(1):8. doi: 10.1186/1710-1492-7-8. PMID 21507261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from advertisement between November 2005 and october 2008
Pre-assignment Details: After enrollment, there was a one to 7 days run-in period. Subjects that could not produce a quality sputum sample were excluded from the trial.
Period: Overall Study
Arm/Group | Allergic Asthmatic | Allergic Rhinitic Without Asthma
Started | 27 | 18
Completed | 19 | 13
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Could not comply with study requirements | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergic Asthmatic | Allergic Rhinitic Without Asthma | Total
Number analyzed (Participants) | 27 | 18 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 18 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (4) | 24 (7) | 24 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 28
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  Canada | 27 | 18 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Sputum Eosinophils Following Allergen Challenge
Description: Eosinophil is an inflammatory cell found in the lungs. Sputum is obtained from hypertonic inhalation. patients expectorate in a sterile dish and mucus plugs are selected and treated to obtain cells. cells are transferred on a slide and a differential count is obtained where eosinophils are counted.
Time Frame: At 7 hours post first and last challenge compared to baseline
Measure: Mean (Standard Error); unit: percentage of sputum eosinophils
Arm/Group | Allergic Asthmatic | Allergic Rhinitic Without Asthma
Number analyzed (Participants) | 19 | 13
percentage of sputum eosinophils
  Baseline percentage eosinophils | 5.6 (1.8) | 2.0 (1.3)
  7h post first challenge percentage eosinophils | 6.0 (1.7) | 1.3 (1.5)
  7h post last challenge percentage eosinophils | 4.1 (1.4) | 1.6 (1.0)

2. Secondary Outcome: Change in Nasal Lavage Eosinophils After Allergen Challenge
Description: Change in nasal lavage eosinophil percentages in allergic asthmatic and allergic non asthmatic at baseline and at 7h post first and last challenge
Time Frame: At 7 hours post first and last challenge compared to baseline
Measure: Mean (Standard Error); unit: percentage of nasal lavage eosinophils
Groups:
- Allergic Asthmatic: Change in nasal lavage eosinophil percentages in allergic asthmatic at baseline and at 7h post first and last challenge
- Allergic Non Asthmatic: Change in nasal lavage eosinophil percentages in allergic non asthmatic at baseline and at 7h post first and last challenge
Arm/Group | Allergic Asthmatic | Allergic Non Asthmatic
Number analyzed (Participants) | 19 | 13
percentage of nasal lavage eosinophils
  Baseline percentage eosinophils | 2.1 (0.6) | 1.3 (0.9)
  7h post first challenge percentage eosinophils | 7.5 (4.3) | 3.0 (1.3)
  7h post last challenge percentage eosinophils | 15.7 (5.4) | 15.5 (9.6)

ADVERSE EVENTS:
Arm/Group | Allergic Asthmatic | Allergic Rhinitic Without Asthma
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/13
Other Adverse Events (participants affected / at risk) | 0/19 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No